CLINICAL TRIAL: NCT01671111
Title: A Phase 2, Open-label, Multicentre, Extension Safety and Tolerability Study for Transfusionally Iron Overloaded Children, Adolescents and Adults Using SSP-004184 (SPD602)
Brief Title: Study for Transfusionally Iron Overloaded Children, Adolescents and Adults Using FBS0701 (SSP-004184)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to treatment stop resulting in an inability to draw conclusions from the data. Evaluation of nonclinical rat findings is ongoing.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD602-301; 2011-006322-25 (EudraCT Number)
Record Dates: First submitted 2012-08-16; First posted 2012-08-23 (Estimated); Results first posted 2015-08-06 (Estimated); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Iron Overload Due to Repeated Red Blood Cell Transfusions

ARMS (1):
- SSP-004814AQ (Experimental)
  Interventions: Drug: SSP-004184AQ

INTERVENTIONS:
Drug: SSP-004184AQ — Long term extension study of 8-75 mg/kg/d of SSP-004184AQ (equivalent to 7-68 mg/kg/d free acid or "active" form)
  Other Names: SPD602

SUMMARY:
The purpose of this extension study is to evaluate SSP-004184AQ in patients with transfusional iron overload and to provide data on long term safety and efficacy.

SSP-004184AQ is an iron chelator under development for chronic daily oral administration to patients with transfusional iron overload

ELIGIBILITY:
Inclusion Criteria:

* Subjects and/or parents willing and able to sign the approved informed consent/and assent (based on institutional guidelines).
* An understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Has either completed a previous SSP-004184AQ study or prematurely discontinued from (with agreement from the Investigator and Shire physician) from one of the SSP-004184AQ studies.
* If applicable, female subjects should be either:

  1. Post-menopausal (12 consecutive months of spontaneous amenorrhea), or
  2. Surgically sterile, or
  3. Females of child-bearing potential must have a negative urine pregnancy test at the Qualification and Enrollment Visit prior to dosing on Day 1. Females of child-bearing potential must agree to abstain from sexual activity that could result in pregnancy or agree to use acceptable methods of contraception.

     For subjects that did not transition directly from their feeder protocol and have initiated treatment with a chelator other than SSP-004184AQ:
* Willing to discontinue all existing iron chelation therapies for a minimum period of 1 to 5 days prior to first dose of SSP-004184AQ.

(Note: This inclusion criterion is also applicable for subjects that were receiving chelators other than SSP-004184AQ in their feeder protocol.)

* Serum ferritin greater than 500 ng/mL at the Qualification and Enrollment Visit.
* Liver iron concentration (LIC) greater than or equal to 2.0 mg iron per g (equivalent dry weight, liver) determined by FerriScan® R2 MRI at the Qualification and Enrollment Visit (Day -28 to Day -8).

(Note: Younger subjects for whom MRI is not feasible will be considered iron overloaded on the basis of serum ferritin only.) - Mean of the previous 3 pre-transfusion hemoglobin concentrations greater than or equal to 7.5 g/dL.

Exclusion:

* Unwilling to remain off all other existing chelation therapies during SSP-004184AQ dosing and for up to 24 hours from last dose.
* A history of non-compliance in a prior FerroKin/Shire-sponsored SSP-004184AQ study (excluding dose suspensions that were medically warranted).
* Cardiac MRI T2* less than 10.0 milliseconds at the Qualification and Enrollment Visit.
* Cardiac left ventricular ejection fraction less than 50% at the Qualification and Enrollment Visit by MRI or below the locally determined normal range by echocardiography if MRI information is not available.
* Evidence of clinically relevant oral, cardiovascular, gastrointestinal, endocrine, pulmonary, neurologic, psychiatric, immunologic, bone marrow, dermatologic, hepatic, biliary, or renal dysfunction where, in the opinion of the Investigator or the Shire Study Physician, treatment with SSP-004184AQ is relatively contraindicated.
* Platelet count below 100,000/µL or absolute neutrophil count less than 1500/mm3 at the Qualification and Enrollment Visit.
* Known sensitivity to any ingredient in the SSP-004184AQ formulation.
* Pregnant or lactating females.

For subjects that did not transition directly from their feeder protocol and have initiated treatment with a chelator other than SSP-004184AQ:

* In younger subjects for whom MRI is not feasible, evidence of severe cardiac dysfunction, as assessed by the Investigator.
* Non-elective hospitalization within the 30 days prior to receiving the first dose of SSP 004184AQ.
* For subjects greater than or equal to 18 years old: ALT greater than 200 IU/L at the Qualification and Enrollment Visit.

OR For subjects less than 18 years old: ALT greater than 180 IU/L at the Qualification and Enrollment Visit.

- For subjects greater than or equal to 18 years old: Evidence of severe renal insufficiency, eg, serum creatinine 1.5X above the upper limit of normal or proteinuria greater than 1 gm per day or a calculated glomerular filtration rate less than 40 mL/min.

OR For subjects less than 18 years old: Evidence of significant renal insufficiency, eg, serum creatinine above the upper limit of normal or proteinuria greater than 1 gm per day.

* Use of any investigational agent within the 30 days prior to receiving the first dose of SSP-004184AQ.
* Cardiac left ventricular ejection fraction below the locally determined normal range in the 12 months prior to Screening by echocardiography or MRI or less than 50% at Baseline testing by MRI (Echocardiograph is acceptable for LVEF if MRI information is not available).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-08-14 (Actual); Primary Completion 2014-04-24 (Actual); Study Completion 2014-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (9):
- United States (2):
  - Children's Hospital Oakland, Oakland, California
  - Children's Hospital of Boston, Boston, Massachusetts
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
- Italy (3):
  - San Luigi Hospital Thalassemia Centre, Orbassano, Torino
  - Ospedale Regionale Microcitemie, Cagliari
  - Ospedale Galliera, Genova
- Siriraj Hospital, Mahidol University, Bangkok, Thailand
- Whittington Hospital, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 30 participants were enrolled to this open-label extension study (24 participants transferred directly from feeder studies SPD602-201 [NCT01186419], SPD602-202 [NCT01363908], and SPD602-203 [NCT01604941] and 6 participants did not transfer directly and received a chelator other than SSP-004184 after discontinuation from a feeder study).
Groups:
- SSP-004184AQ: Participants received SSP-004184AQ (magnesium salt of free acid or active form, that is, SSP-004184 [SPD602, FBS0701]) capsules orally at a total daily dose of 8-75 milligram per kilogram per day (mg/kg/day) (equivalent to SSP-004184 7-68 mg/kg/day) either once daily or twice daily at the discretion of investigator for up to a maximum of 3 years or until the sponsor decided to stop the study.
Period: Overall Study
Arm/Group | SSP-004184AQ
Started | 30
Completed | 0
Not Completed | 30
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1
Not completed — Other | 24

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who had taken at least 1 dose of investigational product.
Groups:
- SSP-004184AQ: Participants received SSP-004184AQ (magnesium salt of free acid or active form, that is, SSP-004184 [SPD602, FBS0701]) capsules orally at a total daily dose of 8-75 mg/kg/day (equivalent to SSP-004184 7-68 mg/kg/day) either once daily or twice daily at the discretion of investigator for up to a maximum of 3 years or until the sponsor decided to stop the study.
Arm/Group | SSP-004184AQ
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ferriscan® R2 Liver Iron Concentrations (LIC) at Week 24 (Cycle 1)
Description: Efficacy of SSP-004184 was assessed by determining LIC. Abdominal magnetic resonance imaging (MRI) data were collected by using FerriScan R2 standard procedures and used to determine LIC. A negative change from baseline indicates that LIC decreased. A cycle consisted of 8 standard 6-weekly visits and the cycles were repeated each year for the duration of the study.
Time Frame: Baseline, Week 24 (Cycle 1)
Population: Full analysis set (FAS) included all participants in the Safety set who had at least 1 post-baseline primary efficacy assessment. Here, 'n' signifies the number of FAS participants evaluable for the respective time points.
Measure: Mean (Standard Deviation); unit: milligram per gram (mg/g) dry tissue
Arm/Group | SSP-004184AQ
Number analyzed (Participants) | 23
milligram per gram (mg/g) dry tissue
  Baseline (n=23) | 9.9 (8.10)
  Change at Week 24 (Cycle 1) (n=13) | -1.1 (1.86)
Statistical Analysis 1: Comparison: SSP-004184AQ; Test type: Superiority or Other; p = 0.0560, paired t-test — P-value was from paired t-test for post treatment timepoint versus baseline

2. Primary Outcome: Change From Baseline in Ferriscan® R2 Liver Iron Concentrations (LIC) at Week 48 (Cycle 1)
Description: Efficacy of SSP-004184 was assessed by determining LIC. Abdominal MRI data were collected by using FerriScan R2 standard procedures and used to determine LIC. A negative change from baseline indicates that LIC decreased. A cycle consisted of 8 standard 6-weekly visits and the cycles were repeated each year for the duration of the study.
Time Frame: Baseline, Week 48 (Cycle 1)
Population: FAS participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: mg/g dry tissue
Arm/Group | SSP-004184AQ
Number analyzed (Participants) | 9
mg/g dry tissue | -1.0 (1.68)
Statistical Analysis 1: Comparison: SSP-004184AQ; Test type: Superiority or Other; p = 0.1232, paired t-test — P-value was from paired t-test for post treatment timepoint versus baseline

3. Primary Outcome: Change From Baseline in Ferriscan® R2 Liver Iron Concentrations (LIC) at Week 24 (Cycle 2)
Description: as for outcome 2
Time Frame: Baseline, Week 24 (Cycle 2)
Population: FAS participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: mg/g dry tissue
Arm/Group | SSP-004184AQ
Number analyzed (Participants) | 7
mg/g dry tissue | -1.5 (2.23)
Statistical Analysis 1: Comparison: SSP-004184AQ; Test type: Superiority or Other; p = 0.1319, paired t-test — P-value was from paired t-test for post treatment timepoint versus baseline

4. Primary Outcome: Change From Baseline in Cardiac T2* Values at Week 24 (Cycle 1)
Description: The efficacy of SSP-004184 was assessed by determining cardiac iron load. Cardiac MRI data were collected by using T2* standard procedures and used to determine iron load. A negative change from baseline indicates that iron load increased. A cycle consisted of 8 standard 6-weekly visits and the cycles were repeated each year for the duration of the study.
Time Frame: Baseline, Week 24 (Cycle 1)
Population: FAS. Here, 'n' signifies the number of FAS participants evaluable for the respective time points.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | SSP-004184AQ
Number analyzed (Participants) | 23
milliseconds
  Baseline (n=23) | 35.14 (12.242)
  Change at Week 24 (Cycle 1) (n=14) | -0.41 (8.069)
Statistical Analysis 1: Comparison: SSP-004184AQ; Test type: Superiority or Other; p = 0.8061, paired t-test — P-value was from paired t-test for log-transformed data at post treatment timepoint versus baseline

5. Primary Outcome: Change From Baseline in Cardiac T2* Values at Week 48 (Cycle 1)
Description: as for outcome 4
Time Frame: Baseline, Week 48 (Cycle 1)
Population: FAS participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | SSP-004184AQ
Number analyzed (Participants) | 9
milliseconds | -3.47 (9.619)
Statistical Analysis 1: Comparison: SSP-004184AQ; Test type: Superiority or Other; p = 0.2297, paired t-test — P-value was from paired t-test for log-transformed data at post treatment timepoint versus baseline

6. Primary Outcome: Change From Baseline in Cardiac T2* Values at Week 24 (Cycle 2)
Description: as for outcome 4
Time Frame: Baseline, Week 24 (Cycle 2)
Population: FAS participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | SSP-004184AQ
Number analyzed (Participants) | 7
milliseconds | -3.91 (5.551)
Statistical Analysis 1: Comparison: SSP-004184AQ; Test type: Superiority or Other; p = 0.1248, paired t-test — P-value was from paired t-test for log-transformed data at post treatment timepoint versus baseline

7. Secondary Outcome: Change From Baseline in Serum Ferritin Values at Specified Visits
Description: A negative change from baseline indicates that serum ferritin decreased. A cycle consisted of 8 standard 6-weekly visits and the cycles were repeated each year for the duration of the study.
Time Frame: Baseline, Weeks 24 and 48 of Cycle 1, Week 24 of Cycle 2
Population: FAS. Here, 'n' signifies the number of FAS participants evaluable for the respective time points.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | SSP-004184AQ
Number analyzed (Participants) | 23
nanogram per milliliter
  Baseline (n=23) | 5353.38 (4588.423)
  Change at Week 24 (Cycle 1) (n=12) | -395.82 (569.305)
  Change at Week 48 (Cycle 1) (n=9) | -250.87 (452.327)
  Change at Week 24 (Cycle 2) (n=7) | -384.03 (649.990)

ADVERSE EVENTS:
Time Frame: From start of study treatment up to the end of study (1 week after the end of treatment)
Description: An adverse event (AE) that occurred during the study was considered a treatment-emergent AE (TEAE) if it had a start date and time on or after the study treatment or if it had a start date before the date and time of the study treatment but increased in intensity on or after the date and time of the study treatment.
Arm/Group | SSP-004184AQ
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 25/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSP-004184AQ (N=30)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSP-004184AQ (N=30)
Influenza like illness (General disorders) | 5 (6)
Nasopharyngitis (Infections and infestations) | 5 (6)
Asthenia (General disorders) | 4 (8)
Nausea (Gastrointestinal disorders) | 4 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Paraesthesia (Nervous system disorders) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Pharyngitis (Infections and infestations) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (3)
Gastroenteritis (Infections and infestations) | 2 (4)
Pyrexia (General disorders) | 2 (5)

LIMITATIONS AND CAVEATS:
This study was terminated early due to non-clinical safety results. Not all participants completed the study. The available efficacy data were analyzed as specified in the statistical analysis plan; however, no efficacy conclusions were drawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.